CLINICAL TRIAL: NCT05113277
Title: Development and Evaluation of a Tonic Immobility Focused Psychoeducational Intervention - Randomized Controlled Trial (RCT)
Brief Title: Development and Evaluation of a Tonic Immobility Focused Psychoeducational Intervention
Acronym: TIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Norman Schmidt, Distinguished Research Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Morabito01
Record Dates: First submitted 2021-09-27; First posted 2021-11-09 (Actual); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-04

CONDITIONS: Posttraumatic Stress Disorder; Tonic Immobility Response
Keywords: Psychoeducation; Online Intervention
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Immobility Response, Tonic

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to complete 1 of 2 interventions - active or control.
Who Masked: Participant
Masking Description: The participant will be randomly assigned to the active or control condition. The participant will not be informed of which condition they are receiving until after completion of the study, at which point individuals in the control condition will be given access to the active intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tonic Immobility Psychoeducation (TIP) (Experimental): Participants in the experimental condition will receive the TIP intervention.
  Interventions: Behavioral: Tonic Immobility Psychoeducation (TIP)
- Health Education Training (HET) (Placebo Comparator): Participants in the control condition will receive the HET intervention.
  Interventions: Behavioral: Health Education Training (HET)

INTERVENTIONS:
Behavioral: Tonic Immobility Psychoeducation (TIP) — TIP is a 45-minute computerized psychoeducation intervention aimed at addressing maladaptive cognitions and emotions associated with TI while using educational and behavioral techniques commonly used in the treatment of trauma-related disorders. Throughout the psychoeducation program vignettes will be presented to clarify concepts and promote participant engagement. In addition, practice exercises and rating scales will be integrated, where applicable, to increase the interactive nature of the program. The following modules will be addressed in the TI psychoeducation intervention: education, myth busting, and behavioral experiments.
  Arms: Tonic Immobility Psychoeducation (TIP)
Behavioral: Health Education Training (HET) — The Healthy Education Training intervention was developed as a 45-minute online intervention that provides education about physical health habits that can impact mental health, such as diet, exercise, and sleep. This intervention has been used in prior clinical trials to control for effects of general education, general coping techniques, and use of technology. Participants in past clinical trials have reported that HET is engaging and beneficial. However, HET is not expected to have an effect on the main symptom outcomes of the current study (guilt, shame, PTSD symptoms).
  Arms: Health Education Training (HET)

SUMMARY:
A randomized controlled trial is planned to evaluate a brief, web-based intervention intended to educate about tonic immobility (TI) within a sample of those who experienced TI in the context of a traumatic event.

DETAILED DESCRIPTION:
A randomized controlled trial is planned to evaluate a brief, web-based intervention intended to educate about tonic immobility (TI) within a sample of those who experienced TI in the context of a traumatic event. The investigators expect that this intervention will lead to improvement in posttraumatic guilt, shame, and PTSD symptoms as compared to an active control condition.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Endorsed prior TI experience (TIQ items A & B)
* Elevated posttraumatic stress symptoms (PCL-5; Blevins et al., 2015)

Exclusion Criteria:

Inability to consent or complete the intervention including:

* Cognitive impairment
* Uncorrected visual or auditory impairment
* Unmedicated severe mental illness
* Imminent risk of harm to self or others

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman B Schmidt, PhD, Principal Investigator — Florida State University
Locations (1):
- Anxiety and Behavioral Health Clinic, Tallahassee, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tonic Immobility Psychoeducation (TIP) | Health Education Training (HET)
Started | 26 | 25
Completed | 18 | 17
Not Completed | 8 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tonic Immobility Psychoeducation (TIP) | Health Education Training (HET) | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.65 (8.90) | 21.48 (5.85) | 22.59 (7.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 23 | 47
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 12 | 15
  Not Hispanic or Latino | 23 | 13 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Participants were instructed to "select all that apply".
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 4 | 0 | 4
    White | 20 | 20 | 40
    More than one race | 0 | 2 | 2
    Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 26 | 25 | 51
Posttraumatic Stress Checklist for DSM-5 [Mean (Standard Deviation); unit: units on a scale] — The posttraumatic stress checklist for DSM-5 (PCL-5) is a 20-item self report measure of posttraumatic stress symptoms. Items are rated from 0 to 4 and totaled for a score ranging between 0 and 80. Higher scores indicated worse symptoms.
  units on a scale | 51.85 (14.15) | 46.6 (16.04) | 49.27 (15.19)
State Shame (State Shame Guilt Scale) [Mean (Standard Deviation); unit: units on a scale] — The State Shame Guilt scale is an 8-item self-report questionnaire with two subscales: state shame and state guilt. Items are rated 1 to 5 and added for a total score of 4 to 20. Higher scores indicate more shame/guilt.
  units on a scale | 9.65 (4.57) | 9.36 (4.83) | 9.51 (4.65)
Posttraumatic Cognitions Inventory [Mean (Standard Deviation); unit: units on a scale] — The Posttraumatic Cognitions Inventory (PTCI) is a 33-item scale designed to assess negative cognitions about the self, negative cognitions about the world, and self-blame occurring post-trauma. Items are rated from 1 to 7 and added for a total score of 33 to 231. Higher scores indicate more problematic posttraumatic cognitions.
  units on a scale | 126.50 (39.09) | 111.38 (36.63) | 119.44 (38.30)
Negative Affect [Mean (Standard Deviation); unit: units on a scale] — Measured using the Positive and Negative Affect Scale, negative affect subscale (PANAS-NA). The PANAS-NA is a 10-item measure of negative affect. Items are rated on a scale form 1 to 5, and added for a total score of 10 to 50 with higher scores indicating more negative affect.
  units on a scale | 25.24 (8.46) | 26.32 (8.13) | 25.78 (8.23)
Anxiety Sensitivity Inventory 3 [Mean (Standard Deviation); unit: units on a scale] — The Anxiety Sensitivity Inventory 3 (ASI-3) is an 18 item self-report questionnaire used to measure fear of anxiety-related symptoms and sensations. Items are rates on a scale from 0 to 4 and added for a total score of 0 to 72, with higher scores indicating higher anxiety sensitivity.
  units on a scale | 35.24 (16.05) | 36.68 (13.85) | 35.96 (14.85)
Life Events Checklist for DSM-5 [Mean (Standard Deviation); unit: Number of items endorsed] — The Life Events Checklist for DSM-5 (LEC-5) is a questionnaire intended to screen for 16 potentially traumatic events that an individual may have experienced, witnessed, and/or learned about in their lifetime. Total number of trauma types experienced, witnessed, and/or learned about is added for a "trauma load" total score ranging between 0 and 48.
  Number of items endorsed | 13.77 (6.94) | 12.6 (5.33) | 13.20 (6.17)
Tonic Immobility Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The Tonic Immobility Questionnaire (TIQ) is a 12-item measures designed to assess tonic immobility experiences across a range of traumatic events. Items are rated on a scale of 0 to 4 for a total score of 0 to 48, with higher scores indicating more severe tonic immobility.
  units on a scale | 32.08 (11.22) | 32.92 (12.03) | 32.49 (11.51)
State Guilt (State Shame Guilt Scale) [Mean (Standard Deviation); unit: units on a scale] — The State Shame Guilt scale is an 8-item self-report questionnaire with two subscales: state shame and state guilt. Items are rated 1 to 5 and added for a total score of 4 to 20. Higher scores indicate more shame/guilt.
  units on a scale | 10.50 (5.03) | 8.40 (4.75) | 9.47 (4.96)

OUTCOME MEASURES:

1. Primary Outcome: Posttraumatic Stress Disorder Symptoms
Description: PTSD symptoms measured using the posttraumatic stress checklist for DSM-5 (PCL-5). The PCL-5 is a 20-item scale with values ranging from 0 to 4 for each item. Items are totaled for a total score ranging 0 to 80, with lower values indicating better outcomes.
Time Frame: up to 1 month
Population: The final sample was comprised of 46 individuals. Of the 51 participants recruited, three participants failed to complete the intervention, as determined at the analysis phase after examining total time spent, and two participants were excluded from analyses due to significantly impairing drug use during the TI experience.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tonic Immobility Psychoeducation (TIP) | Health Education Training (HET)
Number analyzed (Participants) | 25 | 21
units on a scale | 30.41 (18.23) | 31.93 (18.33)

2. Primary Outcome: Guilt
Description: Feelings of guilt as measured using the state shame-guilt scale, 8-item (SSGS-8); Value range = 5 to 20 with lower values indicating better outcomes.
Time Frame: post-intervention, on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tonic Immobility Psychoeducation (TIP) | Health Education Training (HET)
Number analyzed (Participants) | 25 | 21
units on a scale | 6.6 (2.94) | 6.85 (3.86)

3. Primary Outcome: Shame
Description: Feelings of shame as measured using the state shame-guilt scale, 8-item (SSGS-8); Value range = 5 to 20 with lower values indicating better outcomes.
Time Frame: post-intervention, on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tonic Immobility Psychoeducation (TIP) | Health Education Training (HET)
Number analyzed (Participants) | 25 | 21
units on a scale | 6.80 (2.80) | 6.7 (3.76)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored throughout the duration of the study. Each participant was observed from baseline through contacts at baseline, one-week, and one-month follow-up.
Description: No adverse events occurred during the course of the study, to the knowledge of the investigative team. No adverse events were reported by participants to the investigative team or IRB.
Arm/Group | Tonic Immobility Psychoeducation (TIP) | Health Education Training (HET)
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 0/26 | 0/25

LIMITATIONS AND CAVEATS:
Limitations of the study include small sample size and attrition.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-09-27): https://cdn.clinicaltrials.gov/large-docs/77/NCT05113277/Prot_SAP_ICF_000.pdf